CLINICAL TRIAL: NCT03322852
Title: Effect of Clomiphene Citrate on Uterine Hemodynamics in Women With Unexplained Infertility
Brief Title: Effect of Clomiphene Citrate on Uterine Blood Fow in Women With Unexplained Delayed Conception
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eman Omran, principal investigator, Cairo University
Other Study IDs: 4588
Record Dates: First submitted 2017-10-24; First posted 2017-10-26 (Actual); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Vascularization indices observation — The mid-luteal endometrial thickness and volume, uterine vascularization indices of uterine artery pulsatility index and resistance index, endometrial and subendometrial vascularization index, flow index, and vascularization flow index, and serum estradiol and progesterone levels were calculated in spontaneous then stimulated cycles in the same group of infertile patients

SUMMARY:
In a prospective observational study at a university teaching hospital, blood flow indices and serum hormone levels were compared between spontaneous and stimulated cycles in the same group of 50 patients with unexplained delayed conception.

DETAILED DESCRIPTION:
In a prospective observational study at a university teaching hospital, the mid-luteal (peri-implantation) endometrial thickness and volume, uterine artery pulsatility index (PI) and resistance index (RI), endometrial and subendometrial vascularization index, flow index, and vascularization flow index, and serum estradiol and progesterone levels were compared between spontaneous and clomiphene citrate stimulated cycles in the same group of 50 patients with unexplained infertility.

ELIGIBILITY:
Inclusion Criteria:

* Unexplained infertility
* Body mass index less than 30
* Regular menstruation
* Normal pelvic examination and ultrasonography

Exclusion Criteria:

* History of pelvic operations including cesarean section
* History of pelvic inflammatory disease
* Endometriosis
* Pelvic pathology including uterine fibroids
* General disease or medication that could potentially affect pelvic blood flow
* Smoking

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients who had unexplained infertility
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2016-10-01 (Actual); Study Completion 2016-10-30 (Actual)

PRIMARY OUTCOMES:
Flow index of the endometrial region | Day 22 to 24 of the menstrual cycle
  Flow index of the endometrial region was measured by a researcher

SECONDARY OUTCOMES:
Vascularization index of the endometrial region | Day 22 to 24 of the menstrual cycle
  Vascularization index of the endometrial region was measured by a researcher
Vascularization flow index of the endometrial region | Day 22 to 24 of the menstrual cycle
  Vascularization flow index of the endometrial region was measured by a researcher
Vascularization flow index of the sub-endometrial region | Day 22 to 24 of the menstrual cycle
  Vascularization flow index of the sub-endometrial region was measured by a researcher
Flow index of the sub-endometrial region | Day 22 to 24 of the menstrual cycle
  Flow index of the sub-endometrial region was measured by a researcher
Vascularization index of the sub-endometrial region | Day 22 to 24 of the menstrual cycle
  Vascularization index of the sub-endometrial region was measured by a researcher

CONTACTS AND LOCATIONS:
Overall Officials: Eman Omran, M.D., Principal Investigator — Cairo University
Locations (1):
- Department of Obstetrics and Gynecology, Kasr Al-Ainy hospital, Cairo University, Cairo, Greater Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided